CLINICAL TRIAL: NCT03680248
Title: Monitoring of Hepatic Fat Metabolism Using Magnetic Resonance Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Jan Kovar, Head of the laboratory, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: G285
Record Dates: First submitted 2018-09-04; First posted 2018-09-21 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Hepatic Fat Content
Keywords: hepatic fat content; dietary fat; glucose; fructose; non-esterified fatty acid; triglyceride; insulin; postprandial period
MeSH Terms: conditions — Insulin Resistance | interventions — CD36 Antigens; Angptl4 protein, mouse; Glucose; Fructose

STUDY DESIGN:
Intervention Model Description: 10 non-obese insulin-sensitive male volunteers with normal hepatic fat content (less than 5% of liver fat) and 10 non-obese non-diabetic subjects with increased hepatic fat content (more than 5% of hepatic fat) will undergo series of six experiments - changes of liver fat content will be measured at time 0, 3 and 6 hours after specific dietary interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Healthy subjects, Fat (Experimental): non-obese insulin-sensitive male volunteers with normal hepatic fat content (less than 5% of liver fat) - high-fat load intervention
  Interventions: Dietary Supplement: Fat
- Steatosis, Fat (Experimental): non-obese non-diabetic male volunteers with hepatosteatosis (more than 5% of liver fat) - high-fat load intervention
  Interventions: Dietary Supplement: Fat
- Healthy subjects, Fasting (Other): non-obese insulin-sensitive male volunteers with normal hepatic fat content (less than 5% of liver fat) - fasting
  Interventions: Dietary Supplement: Fasting
- Steatosis, Fasting (Other): non-obese non-diabetic male volunteers with hepatosteatosis (more than 5% of liver fat) - fasting
  Interventions: Dietary Supplement: Fasting
- Healthy subjects, Fat+Glucose (Experimental): non-obese insulin-sensitive male volunteers with normal hepatic fat content (less than 5% of liver fat) - high-fat load + glucose administration
  Interventions: Dietary Supplement: Fat+Glucose
- Steatosis, Fat+Glucose (Experimental): non-obese non-diabetic male volunteers with hepatosteatosis (more than 5% of liver fat) - high-fat load + glucose administration
  Interventions: Dietary Supplement: Fat+Glucose
- Healthy subjects, Glucose (Experimental): non-obese insulin-sensitive male volunteers with normal hepatic fat content (less than 5% of liver fat) - glucose administration
  Interventions: Dietary Supplement: Glucose
- Steatosis, Glucose (Experimental): non-obese non-diabetic male volunteers with hepatosteatosis (more than 5% of liver fat) - glucose administration
  Interventions: Dietary Supplement: Glucose
- Healthy subjects, Fat+Fructose (Experimental): non-obese insulin-sensitive male volunteers with normal hepatic fat content (less than 5% of liver fat) - high-fat load + fructose administration
  Interventions: Dietary Supplement: Fat+Fructose
- Steatosis, Fat+Fructose (Experimental): non-obese non-diabetic male volunteers with hepatosteatosis (more than 5% of liver fat) - high-fat load + fructose administration
  Interventions: Dietary Supplement: Fat+Fructose
- Healthy subjects, Fructose (Experimental): non-obese insulin-sensitive male volunteers with normal hepatic fat content (less than 5% of liver fat) - fructose administration
  Interventions: Dietary Supplement: Fructose
- Steatosis, Fructose (Experimental): non-obese non-diabetic male volunteers with hepatosteatosis (more than 5% of liver fat) - fructose administration
  Interventions: Dietary Supplement: Fructose

INTERVENTIONS:
Dietary Supplement: Fat — Subjects will consume dairy cream (150 g of fat) at time 0 hours.
  Arms: Healthy subjects, Fat; Steatosis, Fat
Dietary Supplement: Fasting — Subjects will fast throughout the experiment.
  Arms: Healthy subjects, Fasting; Steatosis, Fasting
Dietary Supplement: Fat+Glucose — Subjects will consume dairy cream (150 g of fat) at time 0 hours. At the same time and 2 and 4 hours later they will drink herbal tea containing 50 g of glucose.
  Arms: Healthy subjects, Fat+Glucose; Steatosis, Fat+Glucose
Dietary Supplement: Glucose — Subjects will drink herbal tea containing 50 g of glucose at times 0, 2 and 4 hours.
  Arms: Healthy subjects, Glucose; Steatosis, Glucose
Dietary Supplement: Fat+Fructose — Subjects will consume dairy cream (150 g of fat) at time 0 hours. At the same time and 2 and 4 hours later they will drink herbal tea containing 50 g of fructose.
  Arms: Healthy subjects, Fat+Fructose; Steatosis, Fat+Fructose
Dietary Supplement: Fructose — Subjects will drink herbal tea containing 50 g of fructose at times 0, 2 and 4 hours.
  Arms: Healthy subjects, Fructose; Steatosis, Fructose

SUMMARY:
The first primary research objective of the study is to determine whether high-fat load (150 g of fat) induces increase in hepatic fat content (HFC) three and six hours after meal in insulin-sensitive subjects with normal HFC (<5% of fat) and in non-diabetic subjects with an increased HFC (>5% of fat). Furthermore, the other objective of the study is to determine whether the response of HFC to a high-fat load is affected by coadministration of glucose or fructose.

DETAILED DESCRIPTION:
The epidemic of non-alcoholic fatty liver disease (NAFLD) is becoming a major challenge faced by health system worldwide. The hepatic fat comes from the major sources - non-esterified fatty acids (NEFA) released from adipose tissue, dietary fat and de novo lipogenesis. Fat accumulation in the liver then occurs when triglycerides (TG) that are formed are not rapidly enough oxidized or secreted from the liver in very low density lipoproteins (VLDL). It can be hypothesized that the capacity of the liver to eliminate TG can be overcome after high load of dietary fat. High-fat load should induce an immediate accumulation of hepatic fat that could be detected using 1H magnetic resonance spectroscopy (1H-MRS). The accumulation of liver fat can be also affected by coadministration of simple carbohydrates - glucose and fructose. The administration of these carbohydrates can have a pronounced impact on the availability of particular sources of hepatic fat.

ELIGIBILITY:
Inclusion Criteria:

* normal response to oral glucose tolerance test
* normal glycated hemoglobin
* normal aspartate aminotransferase (AST)
* normal alanine aminotransferase (ALT)

Exclusion Criteria:

* BMI > 30 kg/m2
* use of pharmacological agents affecting insulin sensitivity
* use of pharmacological agents affecting lipid metabolism
* inability to undergo 1H-MRS examination

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Hepatic fat content | Before time 0 hour, 3 hours, 6 hours
  Change in hepatic fat content as determined by proton magnetic resonance spectroscopy (%) between 0 and 6 hours

SECONDARY OUTCOMES:
TG | before 0, 0.5, 1, 2, 2.5, 3, 4, 4.5, 5, and 6 hours
  Plasma triglyceride concentration
NEFA | before 0, 0.5, 1, 2, 2.5, 3, 4, 4.5, 5, and 6 hours
  Plasma non-esterified fatty-acid concentration
Glucose | before 0, 0.5, 1, 2, 2.5, 3, 4, 4.5, 5, and 6 hours
  Plasma glucose concentration
Insulin | before 0, 0.5, 1, 2, 2.5, 3, 4, 4.5, 5, and 6 hours
  Plasma insulin concentration
Glucagon | before 0, 0.5, 1, 2, 2.5, 3, 4, 4.5, 5, and 6 hours
  Plasma glucagon concentration

CONTACTS AND LOCATIONS:
Overall Officials: Milan Hajek, DSc, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dusilova T, Kovar J, Drobny M, Sedivy P, Dezortova M, Poledne R, Zemankova K, Hajek M. Different acute effects of fructose and glucose administration on hepatic fat content. Am J Clin Nutr. 2019 Jun 1;109(6):1519-1526. doi: 10.1093/ajcn/nqy386. PMID 31136656

DOCUMENTS (2):
  • Study Protocol (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03680248/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03680248/SAP_001.pdf